CLINICAL TRIAL: NCT04802681
Title: Piezo-electric Versus Open Wire Pressure Guidewires for FFR Measurements: Comparison of Two Commercially Available Pressure Wires
Brief Title: Pressure Guidewire Comparison
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lokien van Nunen (Other)
Collaborators: Cavis Technologies AB (Industry)
Responsible Party: Sponsor-Investigator, Lokien van Nunen, Fellow Interventional Cardiology, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PW-COMPARE
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Fractional Flow Reserve; Pressure wire; Drift
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: This study is a prospective single center randomized controlled trial of FFR measurements comparing two commercially available pressure guidewires in consecutive patients undergoing routine FFR measurements in the catheterization laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wirecath - PressureWire X (Other): Patients will undergo simultaneous FFR measurements with the Wirecath and PressureWire X simultaneously.
  Interventions: Device: FFR-measurement with different pressure guidewires

INTERVENTIONS:
Device: FFR-measurement with different pressure guidewires — Measuring FFR with different pressure guidewires

SUMMARY:
Fractional flow reserve (FFR) is the current gold standard for correct decision making with respect to revascularization in the catheterization laboratory. FFR is measured by using a pressure guidewire equipped with a pressure sensor, positioned distal to the stenosis under investigation. A newly developed pressure wire using open wire technology has recently become commercially available. The purpose of this study is to evaluate whether the Wirecath pressure guidewire can be used as standard pressure guidewire.

The effectiveness of the device will be investigated by comparing Wirecath FFR measurements with the measurements of another regular sensor-tipped pressure guidewires during simultaneous FFR measurements in the same vessel.

DETAILED DESCRIPTION:
FFR is a lesion-specific pressure-derived index of functional severity, defined as the maximum myocardial blood flow in the presence of an epicardial stenosis compared with the maximum flow in the hypothetical absence of the stenosis. FFR is measured by advancing a pressure guidewire into the coronary artery distal to the lesion under investigation and maintained in that position. Distal coronary pressure (Pd) and aortic pressure (Pa) are measured simultaneously while inducing steady state maximum hyperemia. FFR is defined as the lowest value of Pd/Pa achieved during maximum hyperemia. An FFR value = or < 0.80 indicates the presence of myocardial ischemia and indicates PCI is warranted.

Existing 0.014" wires with pressure measurement capabilities have been available for more than 20 years. Improvements have been done over time, but they are still regarded as inferior to ordinary guidewires when it comes to maneuverability and general guidewire properties. This is attributed to the microelectronics that are needed to facilitate the pressure measurements in these wires. These existing wires also have issues with signal stability which is often referred to as 'drift'. Drift is an electronical phenomenon that leads to a slow progressive change in the pressure value over time. a not entirely reliable signal quality.

A relatively new pressure guidewire, Wirecath, is an equivalent device to the currently commercially available pressure guidewires. In comparative bench tests it has shown very good maneuverability. Moreover due to the 'open wire' technology (and thus lack of microelectronics throughout the wire), the Wirecath has very stable signal properties and is, according to physical law and bench testing, immune against a hydrostatic error and less affected by drifting of the signal, which are limitations with current pressure guidewires.

This study is designed to examine and compare the pressure measurements of two commercially available pressure guidewires (Abbott and Cavis Technologies) by simultaneously measuring FFR in the same coronary artery with two different pressure guidewires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Scheduled to undergo invasive FFR measurement
* Coronary artery lesions located in the proximal or mid part of the coronary artery
* Reference diameter of at least 2.0mm

Exclusion Criteria:

* Severe aortic valve stenosis
* known conduction disturbances (second- or third-degree AV block)
* acute myocardial infarction (CK >1,000 U/L less than 5 days ago)
* bradycardia (less than 45 beats/min)
* severe hypotension
* extremely tortuous or calcified coronary arteries precluding FFR measurement
* history of severe asthma
* pregnancy
* inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
FFR | During catheterization
  To compare the pressure signals measured by the different available pressure guidewires, specifically the FFR value
Hydrostatic error | During catheterization
  To assess the occurrence of hydrostatic errors when using sensor-tipped wires
Drift | During catheterization
  To assess the occurrence of drift between the different pressure guidewires

SECONDARY OUTCOMES:
Signal quality | During catheterization
  To assess signal quality and stability between the different pressure guidewires
Maneuverability | During catheterization
  To assess maneuverability and handling of the different pressure guidewires

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual (non-anonymized) participant data available to others.

REFERENCES:
- [Derived] Eerdekens R, Tonino PAL, Zimmermann FM, Teeuwen K, Vlaar PJ, de Waard GA, van Royen N, van Nunen LX. Fluid-filled versus sensor-tipped pressure guidewires for FFR and Pd/Pa measurement; PW-COMPARE study. Int J Cardiol. 2024 Jul 1;406:131998. doi: 10.1016/j.ijcard.2024.131998. Epub 2024 Mar 28. PMID 38555057
- [Derived] Ramunddal T, Dworeck C, Torild P, Andreen S, Gan LM, Hirlekar G, Ioanes D, Myredal A, Odenstedt J, Petursson P, Pylova T, Topel F, Volz S, Hilmersson M, Redfors B, Angeras O. Safety and Feasibility Using a Fluid-Filled Wire to Avoid Hydrostatic Errors in Physiological Intracoronary Measurements. Cardiol Res Pract. 2024 Jan 2;2024:6664482. doi: 10.1155/2024/6664482. eCollection 2024. PMID 38204600